CLINICAL TRIAL: NCT06036160
Title: Evaluation de Soins Primaires Intégrés en Psychiatrie
Brief Title: Feasibility of Integrated Care of Depression in Primary Care Pathways
Acronym: ESPRI-PSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association De La Msp Pasteur (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202201
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated care (Experimental)
  Interventions: Other: Integrated care

INTERVENTIONS:
Other: Integrated care — Psychiatric follow-up, cognitive behavioral therapy, physical exercise, psychoeducation

SUMMARY:
This protocol is a feasibility study of an integrated primary care pathway for patients suffering from difficult-to-treat depression. 50 patients will be recruited and followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* Good understanding of french language
* Major depressive disorder based on DSM-V criteria
* MADRS > 19
* FAilure of two antidepressants during 6wks at standard minimal dose

Exclusion Criteria:

* Pregnancy or lactating
* People under tutelage
* bipolar disorder
* no health insurance
* neurological disorders
* contra-indication to physical activity
* high suicidal risk
* first degree history of bipolar disorder, schizophrenia, autism spectrum disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completing the study per-protocol | 3 years

IPD SHARING:
Plan to Share IPD: No